CLINICAL TRIAL: NCT01826097
Title: Non-Invasive Vibrational Device to Improve Sensitivity of Urine Cytology for Bladder Cancer
Brief Title: Improving Sensitivity of Urine Cytology for Bladder Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: NA_00067544
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Bladder Cancer
Keywords: Cytology; Whole body massage vibration
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vibration (Experimental): Whole body vibration applied to a group of 20 bladder cancer patients.
  Interventions: Device: La-Z-Boy Massage Chair Vibration Effect on Bladder Cancer Cell Concentration

INTERVENTIONS:
Device: La-Z-Boy Massage Chair Vibration Effect on Bladder Cancer Cell Concentration

SUMMARY:
Can a commercially available vibrating chair increase the number of urothelial cells in a urine sample of healthy participants non-invasively? The investigators plan is participants will alternate 15 minutes of drinking eight fluid ounces of water and 15 minutes of sitting in the vibrating chair for one hour. The control group will alternate 15 minutes of drinking eight fluid ounces of water and 15 minutes of sitting in a non-vibrating chair for one hour. Then, urine samples will be collected and examined for urothelial cell concentration for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Only adult male subjects who will not have surgery within a period of 2 weeks.
* Over the age of 18
* Have had a confirmed diagnosis of stage 0-4 transitional cell carcinoma within the last 30 days

Exclusion Criteria:

* Cognitive impairment resulting in the inability to give informed consent
* Lack of spoken and written English resulting in the inability to give informed consent
* Presence of infectious disease
* Insulin dependent diabetes mellitus
* Endogenous osteosynthetical material implants
* Knee or hip prosthesis
* Pacemaker
* Epilepsy
* Musculo-skeletal disorders
* Weight in excess of 250 pounds
* Poor circulation

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Cancer Cells | up to 24 weeks
  Number of Cancer Cells in a 50 ml Urine

CONTACTS AND LOCATIONS:
Overall Officials: Trinity Bivalacqua, MD/PhD, Principal Investigator — Johns Hopkins University; John J Kim, BS, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States